CLINICAL TRIAL: NCT06329115
Title: Investigation of the Effectiveness of Regular Physical Activity in University Students Within the Scope of a Course
Brief Title: Investigation of the Effectiveness of Regular Physical Activity in University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assistant Professor, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/23
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Regular Physical Activity; Exercise
Keywords: Physical acitivity; Depression; Anxiety; Sleep quality; Health life learning; Quality of life; Functional capasity; physiological expenditure
MeSH Terms: conditions — Motor Activity; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be included in an 8-week regular exercise program. Evaluations will be made before and after exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Group (Experimental): This group will get aerobic exercise programme and respiratory exercise
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Within the physical activity program, an aerobic training program will be applied to students for a total of 150 minutes per week for 8 weeks. Aerobic training includes moderate-intensity walking exercise. The concept of moderate walking will be explained to individuals at the beginning of the study. Maximal and submaximal heart rate calculations will be made with the formulas (220-age) / (220-age X 0.6) and this heart rate will be maintained throughout the training. Students will have a pedometer application installed on their phones and their step counts and exercise minute data will be recorded. At the same time, in order for students to use their respiratory functions properly during regular walking, diaphragmatic breathing and alternating nose breathing breathing exercises will be taught and they will be instructed to do them once a day with 5 repetitions.

SUMMARY:
In our study, university students who coded the course from various faculties and departments within the scope of a university-wide free elective course, after regular physical activity; It was aimed to examine the effects on lifelong learning, physical activity, fatigue, sleepiness, depression, anxiety and stress levels, quality of life and walking distances and physiological expenditure indices.

DETAILED DESCRIPTION:
Physical activity; They are body movements made using skeletal muscles in daily life and resulting in energy expenditure. In addition to daily living activities such as playing games, doing housework, walking, eating, and bathing, exercise and sports are also included in this definition. Physical activity is very important for a healthy life. Studies have reported that continuing physical activity, especially during growth and young adulthood, has positive effects on aerobic capacity, blood pressure, body composition, glucose metabolism, skeletal health and psychological health. Studies have reported that physical activity affects social and personal success in healthy adult individuals and is associated with sleep quality and depression. In this context, our work; After regular physical activity, university students who code the course from various faculties and departments within the scope of the university-wide free elective course; It was aimed to examine the effects on lifelong learning, physical activity, fatigue, sleepiness, depression, anxiety and stress levels, quality of life and walking distances and physiological expenditure indices.

Hypotheses of the study;

* Regular physical activity improves lifelong learning tendencies in university students.
* Regular physical activity increases the level of physical activity in university students.
* Regular physical activity reduces fatigue levels in university students.
* Regular physical activity reduces daytime sleepiness in university students.
* Regular physical activity improves depression, anxiety and stress levels in university students.
* Regular physical activity improves the quality of life in university students.
* Regular physical activity improves functional capacity and increases walking distance in university students.
* Regular physical activity reduces the physiological expenditure index in university students.

ELIGIBILITY:
Inclusion Criteria:

* Students who choose the course offered within the scope of university-wide elective courses
* No obstacle to aerobic exercise
* No chronic disease
* Individuals who have no history of surgery on the lower extremity in the last 6 months

Exclusion Criteria:

- Individuals who do not volunteer to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Lifelong learning | through of the study, average 8 week
  Lifelong learning processes will be evaluated with the "Lifelong Learning Tendencies Scale" developed by Coşkun in 2009. The 6-point Likert scale (1 = fits a lot, 6 = doesn't fit at all) consists of 27 items and 4 sub-dimensions. It consists of subheadings: Motivation in Lifelong Learning (6 items), Persistence (6 items), Lack of Regulating Learning (6 items), Lack of Curiosity (9 items). The lowest score that can be obtained from the first three dimensions of the scale is 6 (6x1), the middle score (6x3.5) is 21, and the highest score (6x6) is 36. The last dimension, lack of curiosity, was determined as the lowest score (9x1) 9, the middle score (9x3.5) 31.5 and the highest score (9x9) 81 points. In the overall average of the scale, the minimum score that can be obtained from the scale (27x1) is 27, the median score (27x3.5) is 94.5, and the maximum score (27x6) is 162.
Physical activity | through of the study, average 8 week
  International Physical Activity Questionnaire-Short Form (IPAQ) will be used to evaluate physical activity. International Physical Activity Survey Short form (7 questions); It provides information on time spent walking, moderate and vigorous activities, and time spent sitting. Calculation of the total score of the short form includes the sum of the duration (minutes) and frequency (days) of walking, moderate activity and vigorous activity. The energy required for activities is calculated with the MET-minute score. Standard MET values have been established for these activities. Using these values, daily and weekly physical activity levels are calculated.
Fatique | through of the study, average 8 week
  Fatigue levels Gencay et al. It will be evaluated with the "Fatigue Severity Scale", the validity and reliability of which was established in 2012. The scale consists of 9 items. The lowest score that can be achieved among the scale items is 0 and the highest score is 7. As the score increases, the severity of fatigue increases.
Daytime sleepiness | through of the study, average 8 week
  Daytime sleepiness levels of students were developed by John in 1992 and Izci et al. in 2008. It will be evaluated with the "Epworth Sleepiness Scale", whose validity and reliability has been established by. The scale consists of 8 items, the lowest score to be obtained from the scale is 0 and the highest score is 24. As the score increases, the level of daytime sleepiness increases.
Depression, anxiety and stress | through of the study, average 8 week
  Depression, anxiety and stress levels will be evaluated with the "Depression, anxiety and stress scale". The validity and reliability study of the scale was conducted by Sarıçam in 2018. The scale, consisting of 21 items, is scored between 0-3. As the score increases, depression, anxiety and stress levels increase.
Quality of life measurement | through of the study, average 8 week
  The quality of life of students was evaluated by Demiral et al. in 2006. It will be evaluated with the "SF-36 Short Form", whose validity and reliability studies have been conducted by. The survey, which consists of 36 items, includes 8 sub-parameters.Scoring is evaluated separately for each sub-dimension. The total score of the scale is not calculated. In the scale, questions 1, 2 and 11 are about general health, questions 3 are about physical functions, question 4 is about physical role limitation, questions 5 are about emotional role limitation, questions 6 and 10 are about social functions, questions 7 and 8 are about pain, questions 9 are about pain. Statements a, e, g and i of the question question vitality, expressions b, c, d, f and h question mental health. Each subscale is scored between 0 and 100. An increase in the dimension mean score indicates that the quality of life is high in that parameter.
Physiological expenditure indices | through of the study, average 8 week
  The students' resting heart rates and walking heart rates were measured with a pulse oximeter. Physiological expenditure indices will be calculated with the formula = (Heart rate during walking - Resting heart rate) / Walking speed (m/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sallis JF, Prochaska JJ, Taylor WC. A review of correlates of physical activity of children and adolescents. Med Sci Sports Exerc. 2000 May;32(5):963-75. doi: 10.1097/00005768-200005000-00014. PMID 10795788
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Danaei G, Ding EL, Mozaffarian D, Taylor B, Rehm J, Murray CJ, Ezzati M. The preventable causes of death in the United States: comparative risk assessment of dietary, lifestyle, and metabolic risk factors. PLoS Med. 2009 Apr 28;6(4):e1000058. doi: 10.1371/journal.pmed.1000058. Epub 2009 Apr 28. PMID 19399161
- [Background] Booth M. Assessment of physical activity: an international perspective. Res Q Exerc Sport. 2000 Jun;71 Suppl 2:114-20. doi: 10.1080/02701367.2000.11082794. No abstract available. PMID 25680021